CLINICAL TRIAL: NCT05844839
Title: Awareness of Preparatory Schools Girls About Puberty Changes and Menstrual Hygiene in Abnub District
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aml Tharwat Said, resident physician, Assiut University
Other Study IDs: Awareness of menstrual hygiene
Record Dates: First submitted 2023-03-31; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Puberty Changes; Menstrual Hygiene

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
• General objective: Upgrade awareness of adolescent girls during puberty to improve their reproductive health

• Specific objectives:

1. To assess the awareness about pubertal changes and menstrual hygiene among rural and urban adolescent girls.
2. To identify the determinants of awareness about pubertal changes and menstrual hygiene among adolescent girls.
3. To assess the practice of menstrual hygiene among adolescent girls.

DETAILED DESCRIPTION:
Adolescence is one of life's most fascinating and complex stages of human life. The World Health Organization (WHO) defines adolescents as young people aged 10-19 years. Attitudes and behaviors formed in the physical and psychological maturation process are crucial to the current and future Reproductive Health (RH) of individuals, and affect the well-being of their families and communities .

Adolescence is a process-a series of varied, rapid and extensive changes as well as period of life about1/5 of the total female population is contributed by adolescent girls. out of which more than 4/5th residing in developing countries adolescence has challenges that can affect not only the future of a girl but also that of her children .

Reproductive Health is a state of complete physical, mental and social well-being and not merely the absence of disease or infirmity, in all matters relating to the reproductive system, and to its functions and processes. Reproductive health therefore implies that people are able to have a satisfying and safe sex life and that they have the capability to reproduce and the freedom to decide if, when and how often to do so Egypt's young population is rapidly growing. The adolescents (aged 10-19) are around 17 million, representing approximately 19 percent of the total population ,and it is an important stage in the human life span marked by the onset of puberty. It is a stage in which adolescents cross the line between childhood and adulthood Adolescents constitute perhaps the healthiest group in the population, having the lowest mortality and morbidity when compared with other population age groups. Reproductive health covers all aspects of adolescent health. In order to lead healthy, responsible & fulfilling lives & protect themselves from reproductive health problems youngsters need to be knowledge- able about themselves& need adequate information about the physical& psychological changes that take place during puberty, menstruation, pregnancy & child birth Puberty can be a challenging time that is often associated with early sexual activity, dropping out of school, substance abuse, unsuccessful marriage, un- wanted pregnancy, sexually transmitted diseases (STDs) and psychosomatic and social problems Adolescent girls form a group exposed to the possibility of being unsafe not only with respect to their social status but also in relation to their health Puberty mean growth from childhood stage to adolescence stage : This Growth is the result of the concerted effect of a complex network of many regulatory factors with varying interactions In females, the normal start of puberty ranges from 8 to 13 years of age, and it is marked by the development of breast buds under the areola; this step is also called thelarche and represents the Tanner Stage B2. In the sequence of events, the thelarche is followed by pubic and axillary hair growth, known as pubarche; in the meantime, growth velocity starts to increase between stage 2 and 3, reaching a peak in stage 4, when the menarche may appear Menstruation although in natural physiological process often associated with misconceptions and the way a girl gets to know about it can lead to a good or bad perception regarding menstruation. Increased knowledge about menstruation from childhood may increase safe practices and may help in eliminating the suffering of millions of women Inadequate menstrual hygienic practices can harmfully affect the health and can lead to reproductive tract infections, chronic pelvic pain, dysmenorrhea and even infertility The onset of puberty, in addition to the rate of maturation, appears to be dependent on heredity and the environment. The age at menarche of identical twin sisters is within 1-2 months of each other, whereas in dizygotic twins there is about a years difference. In general, girls in poor countries have later menarche than in countries with better socioeconomic conditions .

Age at menarche and breast development are clinically easier to assess, data regarding female puberty is significantly more abundant than male data .

ELIGIBILITY:
Inclusion Criteria:

- Adolescent girls in preparatory schools in Abnub district

Exclusion Criteria:

* Married girls

Ages: 12 Years to 16 Years | Sex: Female
Age Groups: Child
Study Population: Adolescent girls in governmental preparatory schools at Abnub district
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Upgrade awareness of adolescent girls during puberty to improve their reproductive health | 2years
  questionnair will be prepared to assess this outcome